CLINICAL TRIAL: NCT02217579
Title: Effect of Protein and Prebiotic Fiber Intake on Adiposity in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UofC Protocol REB13-0169
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Weight loss; Appetite; Overweight; Obesity; Dietary fiber; Dietary protein
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Isocaloric food without the test protein and prebiotic fiber.
  Interventions: Dietary Supplement: Control
- Protein (Experimental): Dietary protein consumed as two daily servings of 5 grams protein/serving.
  Interventions: Dietary Supplement: Protein
- Fiber (Experimental): Prebiotic fiber consumed as two daily servings of 8 grams protein/serving.
  Interventions: Dietary Supplement: Prebiotic fiber
- Protein plus prebiotic fiber (Experimental): Protein and prebiotic fiber consumed as two daily servings of 5 grams protein/serving plus 8 grams fiber/serving.
  Interventions: Dietary Supplement: Protein plus prebiotic fiber

INTERVENTIONS:
Dietary Supplement: Protein — A food containing 5 grams/serving of supplemental protein.
  Arms: Protein
Dietary Supplement: Prebiotic fiber — A food containing 8 grams/serving of supplemental prebiotic fiber.
  Arms: Fiber
Dietary Supplement: Protein plus prebiotic fiber — A food containing supplemental protein (5 grams/serving) and prebiotic fiber (8 grams/serving).
  Arms: Protein plus prebiotic fiber
Dietary Supplement: Control — An isocaloric food not containing the test protein and fiber.
  Arms: Control

SUMMARY:
The metabolic syndrome is rising worldwide as a consequence of the continued obesity epidemic. The current obesogenic environment makes the regulation of energy intake difficult and impedes the maintenance of weight loss. Dietary patterns and/or ingredients that curb hunger and reduce energy intake are critically needed. We hypothesize that inclusion of protein and prebiotic fiber in the diet will reduce adiposity in overweight and obesity adults.

DETAILED DESCRIPTION:
The main objective of our study is to assess the effects of protein and prebiotic fiber intake on changes in adiposity in an overweight and obese adult population.

Primary objective - To determine the effect of 12 week protein (10 g/day) or prebiotic fiber (16 g/day) intake on changes in body composition, chiefly body fat.

Secondary objective - To measure changes in appetite following 12 weeks of protein (10 g/day) or prebiotic fiber (16 g/day) intake.

Other outcomes includes changes in quality of life ratings and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18 - 70 years
* BMI 25 - 38 kg/m-2
* Stable body weight for at least 3 months prior to the study

Exclusion Criteria:

* Type 1 diabetes
* Clinically significant cardiovascular, liver or pancreas disease
* Major gastrointestinal surgeries
* Pregnant or lactating
* Concomitant use of any weight loss medication, diet or exercise regime
* Antibiotic use in the preceding 3 months to enrollment
* Weight loss > 3 kg within preceding 3 months to enrollment
* Use of bulk laxatives, fiber supplements or probiotic/prebiotic supplements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in baseline fat mass at 12 weeks | 12 weeks
  Assessed with dual energy x-ray absorptiometry.

SECONDARY OUTCOMES:
Change in baseline appetite at 12 weeks | 12 weeks
  Subjective appetite assessed with visual analog scales and objective appetite with a weighed lunch buffet.

OTHER OUTCOMES:
Change in baseline quality of life rating at 12 weeks | 12 weeks
  Measured with SF-36 questionnaire
Change in baseline gut microbiota at 12 weeks | 12 weeks
  Measured by high throughput sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reimer RA, Willis HJ, Tunnicliffe JM, Park H, Madsen KL, Soto-Vaca A. Inulin-type fructans and whey protein both modulate appetite but only fructans alter gut microbiota in adults with overweight/obesity: A randomized controlled trial. Mol Nutr Food Res. 2017 Nov;61(11). doi: 10.1002/mnfr.201700484. Epub 2017 Aug 29. PMID 28730743